CLINICAL TRIAL: NCT05034887
Title: Phase 2 Study of Trastuzumab Deruxtecan in the Neoadjuvant Treatment, or Trastuzumab Deruxtecan Plus Capecitabine Plus Durvalumab(MEDI4736) in the Preoperative and Postoperative Adjuvant Treatment for Patients with HER2 Positive Gastric and Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center Hospital East (Other)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kohei Shitara, Chief of Gastroenterology and Gastrointestinal Oncology Division, National Cancer Center Hospital East
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOC2003
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: Trastuzumab Deruxtecan T-DXd DS-8201a Gastric cancer
MeSH Terms: interventions — trastuzumab deruxtecan; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trastuzumab Deruxtecan (T-DXd) monotherapy (Experimental): One cycle is 21 days, with T-DXd repeated 3 cycles before surgery as the neo adjuvant treatment.
  Interventions: Drug: Trastuzumab Deruxtecan (T-DXd) monotherapy
- Combination cohort (Experimental): T-DXd 5.4 mg/kg and Durvalumab 1500 mg were infused intravenously once 3 weeks, and Capecitabine 750 mg/m2 was administered orally twice daily for 14 days with a 7-day rest period. T-DXd, Capecitabine, and Durvalumab were repeated 3 cycles preoperatively and 3 cycles postoperatively, followed by 10 cycles of Durvalumab monotherapy every 4 weeks.
  Interventions: Drug: T-DXd, Durvalumab and Capecitabine Combination

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan (T-DXd) monotherapy — T-DXd will be administered at a dose of 6.4 mg/kg (decimal) by intravenous infusion every 21 days (3 weeks) for subsequent three cycles.
  Other Names: DS-8201a
  Arms: Trastuzumab Deruxtecan (T-DXd) monotherapy
Drug: T-DXd, Durvalumab and Capecitabine Combination — Administer each cycle over 21 days. T-DXd is administered by intravenous infusion at 5.4 mg/kg every 21 days (every 3 weeks). Capecitabine is given at 750 mg/m2 BID, taken orally for 14 days, followed by a drug holiday from the evening of Day 15 to the morning of Day 22 (Day 1 of the next cycle). Durvalumab is administered at 1500 mg by intravenous infusion over 60 minutes every 21 days (every 3 weeks). As neoadjuvant chemotherapy, administer T-DXd, Capecitabine, and Durvalumab in combination on a q3w schedule for 3 cycles. As adjuvant chemotherapy consists of T-DXd, Capecitabine, and Durvalumab in combination on a q3w schedule for 3 cycles, followed by Durvalumab monotherapy on a q4w schedule until 10 cycles are completed.
  Arms: Combination cohort

SUMMARY:
This study is an open-label, single-arm, multicenter, Phase 2 study to evaluate the efficacy and safety of neoadjuvant chemotherapy with T-DXd monotherapy in patients with HER2-positive gastric cancer.

In the combination cohort, the efficacy and safety of neoadjuvant chemotherapy combined with T-DXd, capecitabine, and durvalumab are evaluated.

DETAILED DESCRIPTION:
This study is an open-label, single-arm, multicenter, phase 2 clinical trial. Eligible patients are with previously untreated gastric and gastroesophageal junction adenocarcinoma as defined by cT2-4 and/or cN+ without evidence of metastatic disease. Study treatment in this study is neoadjuvant treatment with the investigational drug, T-DXd alone, followed by surgery. T-DXd will be administered at a dose of 6.4 mg/kg (decimal) by intravenous infusion every 21 days (3 weeks) for 3 cycles as the neoadjuvant treatment followed by surgery.

In the combination cohort, the efficacy and safety of neoadjuvant chemotherapy combined with T-DXd, capecitabine, and durvalumab are evaluated.

T-DXd 5.4 mg/kg and Durvalumab 1500 mg were infused intravenously once 3 weeks, and Capecitabine 750 mg/m2 was administered orally twice daily for 14 days with a 7-day rest period. T-DXd, Capecitabine, and Durvalumab were repeated 3 cycles preoperatively and 3 cycles postoperatively, followed by 10 cycles of Durvalumab monotherapy every 4 weeks.

Monotherapy will be analyzed in the following 2 analysis sets.

* Patients with HER2 overexpression (IHC3+ or IHC2+ and ISH-positive [FISH or DISH]) in the primary lesion or metastasis (primary analysis part)
* Patients with low expression of HER2 (IHC1+ or IHC2+ and negative for ISH [FISH or DISH]) and HER2-ECD > 11.6 ng/mL in the primary lesion or metastasis (exploratory part)

The combination cohort will be analyzed in the following analysis sets.

- Patients with HER2 overexpression (IHC3+ or IHC2+ and ISH-positive [FISH or DISH]) in the primary lesion or metastasis with gastric adenocarcinoma or GEJ adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the gastric or gastroesophageal junction.
2. Has HER2 overexpression (IHC3+, or IHC2+ and ISH positive [FISH or DISH]). (HER2 Low expression: IHC1+, or IHC2+ and ISH-negative [FISH or DISH] with HER2-ECD > 11.6 ng/mL in the exploratory cohort).
3. Have previously untreated gastric and gastroesophageal junction adenocarcinoma and cT2-4 and/or cN+M0.according to the UICC TNM classification (8th edition),
4. Age ≥ 20 years as the day of informed consent.
5. Has an ECOG performance status (PS) of 0 or 1.
6. Has a left ventricular ejection fraction (LVEF) ≥ 50% by either echocardiogram (ECHO) or multigated collecting acquisition (MUGA) scan within 28 days before enrollment (acceptable on the same day of the week).
7. Has a corrected QT interval (QTc) ≦ 470 ms in females, or QTc ≦ 450 ms in males based on a 12-lead ECG screening within 28 days before enrollment (allowed on the same day of the week). [Fridericia's correction is recommended]
8. Satisfies all of the following requirements within 14 days before enrollment (allowed on the same day of the week).

   * Absolute neutrophil count ≧1500 / mm3 [except for assessment ≦ 14 days after administration of Granules colony-stimulating factors (G-CSF)]
   * Hemoglobin ≧ 8.0 g/dL (except for those measured within 7 days after whole blood transfusion or packed red blood cells)
   * Platelet count ≧100000 per mm3 (excluding measurements within 7 days after platelet transfusion).
   * Total bilirubin ≦1.5 mg/dL (patients with gilbert's syndrome will be allowed if they have < 3.0 mg/dL).
   * AST(GOT)≦100 IU/L
   * ALT(GPT)≦100 IU/L
   * Serum albumin ≧ 2.5 g/dL
   * Calculated creatinine clearance (Cockcroft-Gault ＊) or the actual value ≧ 30 mL/min

     ＊ Cockcroft-Gault equation: creatinine clearance= (140 - age) × body weight (kg) / (72 × Serum creatinine) (* 0.85 x the value obtained for females).
   * PT(INR)< 1.8
   * aPTT < 60 seconds
9. Has a treatment-free period from the end of pre-treatment to before enrollment (allowed on the same day of the week), defined as:

   i. Surgery with general anesthesia : ≧ 4 weeks ii. Radiotherapy: ≧ 4 weeks (including palliative stereotactic body radiation therapy to the chest; palliative stereotactic body radiation therapy to other than the chest ≧ 2 weeks; abdominal vertebral bodies should be included in the abdomen).

   iii. Chloroquine and hydroxychloroquine : ≧ 15 days
10. Has a prior radiotherapy or surgical AE recovered of ≦ Grade 1 or ≦ baseline on CTCAE v5.0. However, this shall not apply to events where the symptoms are stable even if they are grade 2 or higher.
11. Female of childbearing potential have a negative pregnancy test within 7 days before enrollment (allowed on the same day of the week). Male and Female of childbearing potential agree to contraception for a period (4 months for male and 7 months for Female) from informed consent to the last dose of study drug (see 4.3 "Pregnancy and contraception").
12. Written informed consent of participation in the study has been obtained from the patient.

Exclusion Criteria:

1. Has a medical history of myocardial infarction or congestive heart failure (New York Heart Association Classes II-IV) within 6 months before enrollment, corresponding to the value diagnosed as myocardial infarction as defined by the *validated test within 28 days before enrollment (allowed on the same day), unstable angina, or any serious arrhythmia requiring treatment.

   * tested in local institutions **: Enrollment is allowed with value exceeds ULN if myocardial infarction can be excluded.
2. Active other cancers [Synchronous other cancers and metachronous other cancers within 3 years prior to enrollment, but carcinoma in situ or other lesions corresponding to mucosal carcinoma that are considered curable with local treatment will not be included in active other cancers.]
3. Has serious (hospitalized) complications (intestinal palsy, intestinal obstruction, pulmonary fibrosis, diabetes mellitus that is difficult to control, heart failure, myocardial infarction, unstable angina, renal failure, liver failure, psychiatric disorders, cerebrovascular disorders, etc.).
4. Has history of gastrointestinal perforation and/or gastrointestinal fistula within 6 months before enrollment.
5. Has any of the following infections:

   * HBs antigen positive
   * HBs antibody or HBc antibody and HBV-DNA positive
   * Active hepatitis C (eg, if HCV RNA is detected qualitatively) Patients who are HBsAg positive but who have achieved HBV DNA level < 1.3 log IU/mL (2.1 log copies/mL) after treatment with antiviral drugs such as NAs, are eligible for the study.
6. HIV infection
7. Lung diseases defined as:

   * Has a history of non-infectious interstitial lung disease or pneumonitis that required treatment, has interstitial lung disease or pneumonitis, or these lung diseases cannot be ruled out by radiographic examination before enrollment.
   * Severe pulmonary disease (eg, pulmonary embolism within 3 months prior to enrollment, serious bronchial asthma, severe COPD, restrictive pulmonary disease, or pleural effusion).

   Lung-related autoimmune or connective tissue or inflammatory diseases (eg, rheumatoid arthritis, Sjögren's syndrome, or sarcoidosis) with clinically severe pulmonary risks.

   • Has history of pneumonectomy.
8. Has history of concomitant autoimmune disease or chronic or recurrent autoimmune disease.
9. Administration of systemic corticosteroids (except prophylactic administration for diagnostic tests or allergic reactions, and temporary use for the purpose of reducing edema associated with radiotherapy) or immunosuppressants is required, or has received these treatments within 14 days before enrollment in the study.
10. Has unhealed wounds, ulcers, or fractures.
11. If patients are a pregnancy or breastfeeding patient.
12. Has documented severe hypersensitivity to study drug active ingredients or additives.
13. Has history/complications of severe hypersensitivity reactions to other monoclonal antibodies.
14. has uncontrolled acute systemic infection that requires Infusion intravenous antibiotic, antiviral, or antifungal drug.
15. Unwilling or unable to follow study protocol or any of the instructions by the physician.
16. The investigator or subinvestigator considered it ineligible for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Major pathological response [MPR] rate: by central assessment | 6 months
  MPR is defined as the proportion of subjects with < 10% residual tumor in the stomach and lymph nodes by central assessment

SECONDARY OUTCOMES:
MPR rate determined by the local assessment | 6 months
  The proportion of subjects with MPR by Local assessment
Pathological complete response (pCR) rate | 6 months
  The proportion of subjects with complete remission of gastric and lymph node tumors by local assessment
Curative Resection Rate | 6 months
  Defined as the proportion of subjects who start study treatment and undergo radical resection (R0)
AE rate | From the start day of study treatment, "47 days after the last dose, 30 days after surgery, or if postoperative adjuvant chemotherapy or treatment is started before it, whichever comes first.
  The treatment-emergent AEs will be summarized by CTCAE v5.0.
Percentage of completed treatment before surgery (Combination cohort only) | 3 years
  The proportion of subjects who underwent radical resection (R0) after the initiation of the study treatment and the completion of the 3 cycles of the study treatment is defined as the proportion of subjects who underwent radical resection (R0).
Percentage of completed postoperative adjuvant chemotherapy (Combination cohort only) | 3 years
  The proportion of subjects who received 3 cycles of the study drug until radical resection (R0) and received 13 cycles of adjuvant chemotherapy after the initiation of the study treatment.
Event-Free Survival (EFS) (Combination cohort only) | 3 years
  The date of registration is defined as the start date and the time to the event that occurred whichever comes first:
  * Disease progression based on imaging evaluations using RECIST 1.1
  * Local or distant recurrence based on CT or biopsy in patients without postoperative lesions
  * Death from any cause
Overall Survival (OS) (Combination cohort only) | 3 years
  The date of registration is defined as the start date and the time to death from any cause is defined as the period from the start date of registration.

OTHER OUTCOMES:
Biomarkers in the Primary cohort and the Exploration cohort | 6 months
  Change of ctDNA and examination of various biomarkers.
MPR rate determined by investigator assessment in the Exploration cohort | 6 months
  The proportion of subjects with< 10% residual tumor in the stomach and lymph nodes
pCR rate determined by investigator assessment in the Exploration cohort | 6 months
  The proportion of subjects with complete remission of gastric and lymph node tumors
Curative Resection Rate in the Exploration Part | 6 months
  Defined as the proportion of subjects who start study treatment and undergo radical resection (R0).
AE rate in the Exploration Part | From the start day of study treatment, "47 days after the last dose, 30 days after surgery, or if postoperative adjuvant chemotherapy or treatment is started before it, whichever comes first.
  The treatment-emergent AEs will be summarized by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Kohei Shitara, MD, Principal Investigator — National Cancer Center Hospital East
Locations (1):
- National Cancer Center Hospital East, Kashiwa, Chiba, Japan

IPD SHARING:
Plan to Share IPD: No